CLINICAL TRIAL: NCT00004867
Title: The Utility of Positron Emission Tomography (PET) in Staging of Patients With Potentially Operable Carcinoma of the Thoracic Esophagus
Brief Title: Positron Emission Tomography in Determining Stage of Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACOSOG-Z0060; CDR0000067526 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Esophageal Cancer
Keywords: stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18; Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FDG-PET scan +/- neoadjuvant chemotherapy + surgery (Experimental): Patients receive fludeoxyglucose F 18 (FDG) IV followed 45-60 minutes later by positron emission tomography (PET) imaging. Confirmatory studies, such as biopsy or other imaging studies, are then conducted to confirm the FDG PET imaging results. Patients with no metastases identified by FDG PET imaging may undergo esophagectomy with or without neoadjuvant chemoradiotherapy within 1 month of evaluation.
  Patients are followed within 6 months after surgery.
  Interventions: Procedure: conventional surgery; Procedure: positron emission tomography; Procedure: radionuclide imaging; Radiation: fludeoxyglucose F 18; Drug: chemotherapy; Radiation: Radiotherapy

INTERVENTIONS:
Procedure: conventional surgery
Procedure: positron emission tomography
Procedure: radionuclide imaging
Radiation: fludeoxyglucose F 18
Drug: chemotherapy
Radiation: Radiotherapy

SUMMARY:
RATIONALE: Imaging procedures such as positron emission tomography may improve the ability to determine the stage of esophageal cancer.

PURPOSE: This clinical trial is studying how well fludeoxyglucose F 18 positron emission tomography determines tumor stage in patients with esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objective:

To evaluate whether FDG-PET imaging can detect lesions that would preclude surgery (esophagectomy) in patients found to be surgical candidates by standard imaging procedures.

Secondary Objective:

To use the collected data to generate hypotheses to be used in future studies, such as which types of previously undetected lesions FDG-PET imaging is best able to identify.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be ≥ 18 years of age.
2. Patient must have histologically confirmed squamous cell carcinoma or adenocarcinoma of the thoracic esophagus (greater than or equal to 20 cm from incisors) or gastroesophageal junction. (Pathology report must be submitted).
3. Patient must be deemed medically fit for surgical staging procedures and esophagectomy following the thoracic surgeon's evaluation of general medical fitness.
4. Patient's clinical staging data (clinical examination, laboratory tests, and standard radiological staging assessments) must be obtained within 60 days prior to registration and must suggest that the tumor is potentially resectable, including tumors staged T1-3, N0-1, M0.
5. Patient must be able to tolerate FDG-PET scan (e.g., not claustrophobic and able to lie supine for 1.5 hrs).
6. Female patient of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to FDG-PET.

   * NOTE: Pregnancy test is required to avoid unnecessary fetal radiation exposure and because the use of furosemide is contraindicated in pregnancy.
7. Patient or the patient's legally acceptable representative must provide a signed and dated written informed consent prior to registration and any study related procedures.
8. Patient must provide written authorization to allow the use and disclosure of their protected health information.

   * NOTE: This may be obtained in either the study-specific informed consent or in a separate authorization form and must be obtained from the patient prior to study pre-registration.
9. A cancer survivor is eligible provided that ALL of the following criteria are met and documented:

   * the patient has undergone potentially curative therapy for all prior malignancies and
   * there has been no evidence of any prior malignancies for at least five years (except for completely resected cervical or non-melanoma skin cancer) and
   * the patient is deemed by their treating physician to be at low risk for recurrence from prior malignancies.

Exclusion Criteria:

1. Patient has proximal esophageal cancer (less than 20 cm from incisors) potentially requiring pharyngolaryngoesophagectomy.
2. Patient has unresectable lesions (stage M1b, with biopsy confirmation of distant metastatic disease; or those with unresectable locoregional invasion, T4 Nx Mx).
3. Patient has evidence of metastatic disease.

   * NOTE: Obvious metastasis that is based on clinical evaluation includes any or all of the following: positive cytology of pleura, pericardium, or peritoneum; metastasis to brain, bone, lung, liver, or adrenals; positive biopsy or cytology of metastasis to supraclavicular lymph nodes; and involvement of the tracheobronchial tree (positive bronchoscopic biopsy or overt esophago-respiratory fistula).
4. Patient has had a prior FDG-PET scan for evaluation of their esophageal cancer.
5. Patient has uncontrolled diabetes mellitus, as evidenced by a fasting blood glucose value >200 mg/dL, within 12 hours of FDG-PET scan.
6. Patient has received neoadjuvant chemotherapy and/or radiotherapy PRIOR to FDG-PET scan being performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 1999-11; Primary Completion 2005-07 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Proportion of these patients with FDG-PET findings that contraindicate surgery | Up to 1 month post-FDG-PET scan

SECONDARY OUTCOMES:
The proportion of false positive lesions found by FDG-PET. | Up to 6 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bryan F. Meyers, MD, MPH, Study Chair — Washington University Siteman Cancer Center
Locations (35):
- United States (35):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - University of South Alabama Cancer Research Institute, Mobile, Alabama
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Morton Plant Hospital, Clearwater, Florida
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Cancer Center at Greater Baltimore Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Tri-Health Good Samaritan Hospital, Cincinnati, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Westmoreland Regional Hospital, Greensburg, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - St. Clair Memorial Hospital, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis, Memphis, Tennessee
  - Veterans Affairs Medical Center - Tennessee Valley Healthcare System - Nashville Campus, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington

REFERENCES:
- [Result] Veeramachaneni NK, Zoole JB, Decker PA, Putnam JB Jr, Meyers BF; American College of Surgeons Oncology Group Z0060 Trial. Lymph node analysis in esophageal resection: American College of Surgeons Oncology Group Z0060 trial. Ann Thorac Surg. 2008 Aug;86(2):418-21; discussion 421. doi: 10.1016/j.athoracsur.2008.04.043. PMID 18640307